CLINICAL TRIAL: NCT03471143
Title: Phase 1/2a Study of 2-Hydroxypropyl-Beta-Cyclodextrin Therapy for Infantile Liver Disease Associated With Niemann-Pick Disease, Type C
Brief Title: Study of IV VTS-270 for Infantile Liver Disease Associated With Niemann-Pick Disease, Type C
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201708114; 5U01HD090845-04 (NIH)
Record Dates: First submitted 2018-03-07; First posted 2018-03-20 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Niemann-Pick Disease, Type C
MeSH Terms: conditions — Niemann-Pick Disease, Type C | interventions — 2-Hydroxypropyl-beta-cyclodextrin

STUDY DESIGN:
Intervention Model Description: Phase 1/2a, open-label, dose escalation, multi-center study of adrabetadex (VTS-270) in subjects with NPC dosed twice a week with IV adrabetadex (VTS-270) for six weeks for a total of 12 administrations, followed by a six month open-label extension phase in which the subjects are dosed monthly with IV adrabetadex (VTS-270) for six months for a total of six administrations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IV adrabetadex (VTS-270) for NPC1 infants (Experimental): Phase 1: Dosing frequency will be twice a week administered via a peripherally inserted central catheter (PICC) for six weeks for a total of 12 administrations. Doses 3-12 will occur as an outpatient.
  Doses to be studied are 500, and 1000 mg/kg. Six subjects will be studied at each dose level. Cohort 1: Subjects 1-6 will receive 500 mg/kg Cohort 2: Subjects 7-12 will receive 1000 mg/kg Subjects who demonstrate significant reduction either in the glycine-conjugated trihydroxycholanic acid biomarker or serum bilirubin (direct bilirubin or direct bilirubin:total bilirubin ratio) will be allowed to crossover into the second phase of the study, an open-label phase of six months duration. In the this phase of the study, dosing frequency will be monthly with IV VTS-270 administered via peripheral IV access for six months for a total of six administrations.
  Interventions: Drug: VTS-270

INTERVENTIONS:
Drug: VTS-270 — VTS-270 (2-Hydroxypropyl-Beta-Cyclodextrin) will be administered intravenously to specifically target liver disease. In the first phase of the study, dosing frequency will be twice a week with IV adrabetadex (VTS-270) for six weeks for a total of 12 administrations. Subjects will be evaluated at each study visit for evidence of adverse effects.
  Doses to be studied are 500, and 1000 mg/kg. Six subjects will be studied at each dose level. Cohort 1: Subjects 1-6, 500 mg/kg Cohort 2: Subjects 7-12, 1000 mg/kg
  Other Names: adrabetadex

SUMMARY:
Niemann-Pick disease, type C (NPC) is a lethal, autosomal recessive, lysosomal storage disorder characterized by neurodegeneration in early childhood and death in adolescence. NPC results from mutation of either the Niemann-Pick C1 disease (NPC1) (~95% of cases) or NPC2 genes. NPC is characterized by the endolysosomal storage of unesterified cholesterol and lipids in both the central nervous system and peripheral tissues such as the liver. Individuals with NPC demonstrate progressive central nervous system decline including inability to coordinate balance, gait, extremity and eye movements. Acute liver disease in the newborn/infant period is frequently observed, but subsequently resolves. However, chronic, sub-clinical liver disease persists. Intrathecal 2-Hydroxypropyl-β-Cyclodextrin (HP-β-CD, VTS-270), also known as adrabetadex, has proven effective in reducing the signs and prolonging life in animal models and Phase 1/2a data support efficacy in NPC1 patients. Adrabetadex (VTS-270) also has been shown to be effective in treating liver disease in the NPC1 cat.

This Phase 1/2a, open-label, multiple ascending dose trial will evaluate whether adrabetadex (VTS-270) administered intravenously is effective in treating acute liver disease in NPC1 infants.

DETAILED DESCRIPTION:
In the first phase of the study, infants will be treated for a total of 6 weeks, treated twice weekly. Infants will be admitted to the Neonatal Intensive Care Unit (NICU) for the first week of treatment. Procedures during the first week of the study will include blood draws for genetic testing, clinical and research blood draws, urine collection, abdominal ultrasound, peripheral inserted central catheter (PICC) placement, hearing screening, and the first two IV adrabetadex (VTS-270) infusions through the PICC line. Weeks 2-6 will occur on an outpatient basis. During week 2-6, the infant will receive 2 doses per week of adrabetadex (VTS-270) with blood draws and urine collection during weeks 2, 4, and 6. PICC line will be removed after final infusion.

Subjects who demonstrate significant reduction either in the glycine-conjugated trihydroxycholanic acid biomarker or serum bilirubin (direct bilirubin or direct bilirubin: total bilirubin ratio) will be allowed to crossover into the second phase of the study, an open label phase of six months duration in which IV adrabetadex (VTS-270) will be administered monthly for a total of six doses. Month 1-6 procedures will occur on an outpatient basis. Procedures during the second phase include a monthly intravenous line placement. After each monthly visit, the intravenous line will be removed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0 to 6 months of age at time of enrollment, both genders, and any race/ethnicity.
2. Diagnosis of NPC (either NPC1 or NPC2) based upon meeting any of the two following conditions:

   A. Two variants classified as pathogenic or likely pathogenic in NPC1/NPC2 on clinical laboratory testing, or B. One variant classified as pathogenic or likely pathogenic on clinical laboratory testing and a positive NPC biochemical marker (oxysterol or bile acid biomarker or PPCS/Lyso509) test, if acid sphingomyelinase deficiency and cholesterol ester storage disease have been excluded either by clinical molecular testing of the SMPD1 and LIPA genes or by clinical biochemical assay for acid sphingomyelinase and lysosomal acid lipase enzymes (or a combination of enzymatic and molecular testing).

   Variants will be interpreted using the American College of Medical Genetics guidelines for the interpretation of sequence variants (2015) and testing must be performed by a CLIA-certified laboratory.
3. Subjects with evidence of NPC-related liver disease as defined by direct bilirubin (DB) >2mg/dL or DB/total bilirubin ratio >0.2.
4. Ability to travel to a research site.
5. Willing to participate in all aspects of trial design including serial blood collections.
6. Parent / guardian must provide written informed consent to participate in the study. Because of the age range intended for inclusion, assent will not possible.

Exclusion Criteria:

1. Age > 6 months at time of enrollment in the trial.
2. A medical condition (such as clinically significant bleeding diathesis or evidence of immune suppression) that in the opinion of the investigator precludes placement of an intravenous catheter
3. An absolute neutrophil count (ANC) of less than 1,500 per microliter.
4. A platelet count less than 75,000 per microliter.
5. History of severe neonatal encephalopathy, per modified Sarnat including level of consciousness as stupor/coma, absent spontaneous activity, decerebrate posture, flaccid tone, absent suck, absent moro, diverted/nonreactive pupils, lack of heart rate variability, apnea.
6. Subjects, who in the opinion of the investigators, are unable to comply with the protocol or have specific health concerns that would potentially increase the risk of participation. Examples of inability to comply include unwillingness to relocate or travel to a study site, suspected noncompliance with study procedures, behavior that jeopardizes the safety or security of the data or study staff, and other causes of inability to comply.
7. Concurrent participation in another investigational drug trial.
8. History of renal disease or evidence of acute kidney injury defined as serum creatinine greater than 1.5 mg/dL or an increase of at least 0.2-0.3 mg/dL per day.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia I Dickson, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ory DS, Ottinger EA, Farhat NY, King KA, Jiang X, Weissfeld L, Berry-Kravis E, Davidson CD, Bianconi S, Keener LA, Rao R, Soldatos A, Sidhu R, Walters KA, Xu X, Thurm A, Solomon B, Pavan WJ, Machielse BN, Kao M, Silber SA, McKew JC, Brewer CC, Vite CH, Walkley SU, Austin CP, Porter FD. Intrathecal 2-hydroxypropyl-beta-cyclodextrin decreases neurological disease progression in Niemann-Pick disease, type C1: a non-randomised, open-label, phase 1-2 trial. Lancet. 2017 Oct 14;390(10104):1758-1768. doi: 10.1016/S0140-6736(17)31465-4. Epub 2017 Aug 10. PMID 28803710

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The original enrollment goal was 12 subjects up to maximum of 15 subjects to account for potential study withdrawals, discontinuations or unconfirmed diagnosis of NPC.
  Six subjects would be studied at each dose level. Cohort 1: Subjects 1-6 500mg/kg Cohort 2: Subjects 7-12 1000mg/kg
  The four subjects enrolled received 500mg/kg study drug.
Groups:
- IV Adrabetadex (VTS-270) for NPC1 Infants: Treatment group dosing was 500mg intravenous adrabetatex twice a week for 6 weeks, then received 500mg intravenous adrabetatex monthly for 6 months.
Period: Overall Study
Arm/Group | IV Adrabetadex (VTS-270) for NPC1 Infants
Started | 4
Completed | 3
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- IV Adrabetadex (VTS-270) for NPC1 Infants: IV Adrabetadex (VTS-270) for NPC1 Infants. Will measure plasma level of 5α-cholanic acid-3β, 5α, 6β-triol N-(carboxymethyl)-amide.
Arm/Group | IV Adrabetadex (VTS-270) for NPC1 Infants
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Plasma level of 5α-cholanic acid-3β, 5α, 6β-triol N-(carboxymethyl)-amide [Median (Inter-Quartile Range); unit: ng/ml] — Plasma levels of 5α-cholanic acid-3β, 5α, 6β-triol N-(carboxymethyl)-amide will be measured in ng/ml from blood drawn from the participants at baseline.
  ng/ml | 120.6 [96.2 to 145]
Aspartate aminotransferase (AST) [Median (Inter-Quartile Range); unit: U/L] | 168 [167 to 169]
Alanine transaminase (ALT) [Median (Inter-Quartile Range); unit: U/L] | 158.5 [124 to 193]
Spleen volume [Median (Inter-Quartile Range); unit: cc] | 86.3 [84.2 to 88.4]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Adrabetadex (VTS-270) to Reduce Plasma Levels of a Conjugated Bile Acid, Known as 5α-cholanic Acid-3β, 5α, 6β-triol N-(Carboxymethyl)-Amide
Description: This bile acid, 5α-cholanic acid-3β, 5α, 6β-triol N-(carboxymethyl)-amide, is elevated >99% of NPC1 subjects, is largely generated in the liver and therefore provides a biochemical measure of oxidizable lysosomal unesterified cholesterol in liver tissue. The primary outcome measure in phase 1 of the study is the change in plasma levels of 5α-cholanic acid-3β, 5α, 6β-triol N-(carboxymethyl)-amide measured in nanograms/ml from baseline to 6 weeks. The primary outcome measure in phase 2 of the study is the change in plasma levels of 5α-cholanic acid-3β, 5α, 6β-triol N-(carboxymethyl)-amide measured in nanograms/ml from 6 weeks to the end of the 6 month treatment period.
Time Frame: Phase 1: 6 weeks; Phase 2: 6 months
Population: One of the participants only had baseline measurement.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Groups:
- IV Adrabetadex (VTS-270) for NPC1 Infants: In this Phase 1/2a open label trial, there was only 1 arm for treatment, with no comparison group. There was no dose escalation. All participants received 500 mg/kg.adrabetadex (2-Hydroxypropyl-Beta-Cyclodextrin). In Phase 1: Dosing frequency was twice a week administered via a peripherally inserted central catheter (PICC) for six weeks up to a total of 12 administrations.
  Subjects who demonstrated significant reduction either in the glycine-conjugated trihydroxycholanic acid biomarker or serum bilirubin (direct bilirubin or direct bilirubin:total bilirubin ratio) were allowed to crossover into the second phase of the study, an open-label phase of six months duration. In the this phase of the study, dosing frequency was monthly with IV VTS-270 administered via peripheral IV access for six months for a total of six administrations.
Arm/Group | IV Adrabetadex (VTS-270) for NPC1 Infants
Number analyzed (Participants) | 3
ng/ml
  6 weeks | 32.6 [10.5 to 129]
  6 months | 87.9 [46.6 to 101]

2. Secondary Outcome: Effect of Drug on Serum Transaminases
Description: Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) are elevated with liver dysfunction. The outcome measure in phase 1 of the study is the change in ALT and AST levels from baseline to 6 weeks. The outcome measure in phase 2 of the study is the change in ALT and AST levels from 6 weeks to the end of the 6 month treatment period.
Time Frame: Phase 1: 6 weeks; Phase 2: 6 months
Population: One of the participants only had baseline measurement.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | IV Adrabetadex (VTS-270) for NPC1 Infants
Number analyzed (Participants) | 3
U/L
  ALT 6 weeks | 87 [80 to 203]
  AST 6 weeks | 114 [86 to 293]
  ALT 6 months | 65 [48 to 71]
  AST 6 months | 77 [75 to 89]

3. Secondary Outcome: Reduction of Liver and/or Spleen Volumes
Description: Abdominal ultrasound. The outcome measure in phase 1 of the study is the change in liver and/or spleen volumes from baseline to 6 weeks. The outcome measure in phase 2 of the study is the change in liver and/or spleen volumes from 6 weeks to the end of the 6 month treatment period.
  We were only able to collect spleen volume data due to the radiologist reporting they could not accurately obtain liver volume data. The contact radiologist for this protocol has left the institution, stopping any additional work on liver ultrasound volumes. None of the remaining radiology colleagues had time to bring forward. Liver volumes will never be obtained for this measure in the future.
Time Frame: Phase 1: 6 weeks; Phase 2: 6 months
Population: We were only able to collect spleen volume data due to the radiologist reporting they could not accurately obtain liver volume data. The contact radiologist for this protocol has left the institution, stopping any additional work on liver ultrasound volumes. None of the remaining radiology colleagues had time to bring forward. Liver volumes will never be obtained for this measure in the future.
Measure: Median (Inter-Quartile Range); unit: cc
Groups:
- Treatment Group: Treatment group only, no comparison.
  .
Arm/Group | Treatment Group
Number analyzed (Participants) | 3
cc
  6 weeks | 71.8 [58.6 to 98.1]
  6 months | 127 [69.2 to 177.2]

ADVERSE EVENTS:
Time Frame: 7 months and 2 weeks
Groups:
- IV Adrabetadex (VTS-270) for NPC1 Infants: Phase 1: Dosing frequency will be twice a week administered via a peripherally inserted central catheter (PICC) for six weeks for a total of 12 administrations. Doses 3-12 will occur as an outpatient.
  Doses to be studied are 500, and 1000 mg/kg. Six subjects will be studied at each dose level. Cohort 1: Subjects 1-6 will receive 500 mg/kg Cohort 2: Subjects 7-12 will receive 1000 mg/kg Subjects who demonstrate significant reduction either in the glycine-conjugated trihydroxycholanic acid biomarker or serum bilirubin (direct bilirubin or direct bilirubin:total bilirubin ratio) will be allowed to crossover into the second phase of the study, an open-label phase of six months duration. In the this phase of the study, dosing frequency will be monthly with IV VTS-270 administered via peripheral IV access for six months for a total of six administrations.
  adrabetadex (2-Hydroxypropyl-Beta-Cyclodextrin): VTS-270 (2-Hydroxypropyl-Beta-Cyclodextrin) will be administered intravenously to specifically target liver disease. In the first phase of the study, dosing frequency will be twice a week with IV adrabetadex (VTS-270) for six weeks for a total of 12 administrations. Subjects will be evaluated at each study visit for evidence of adverse effects.
  Doses to be studied are 500, and 1000 mg/kg. Six subjects will be studied at each dose level. Cohort 1: Subjects 1-6, 500 mg/kg Cohort 2: Subjects 7-12, 1000 mg/kg
Arm/Group | IV Adrabetadex (VTS-270) for NPC1 Infants
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Adrabetadex (VTS-270) for NPC1 Infants (N=4)
Death (Hepatobiliary disorders) | 1 (1)
Hospitalization (Infections and infestations) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Adrabetadex (VTS-270) for NPC1 Infants (N=4)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
limited vertical gaze (Eye disorders) | 1 (1)
small umbilical hernia (General disorders) | 2 (2)
1/6 systolic murmur (Cardiac disorders) | 1 (1)
dry skin and maculopapular rash on both cheeks (Skin and subcutaneous tissue disorders) | 1 (1)
elevated prothrombin time (Hepatobiliary disorders) | 2 (2)
diaper rash (Skin and subcutaneous tissue disorders) | 1 (1)
right ventricular hypertrophy on ECG (Cardiac disorders) | 1 (1)
mild truncal hypotonia (Nervous system disorders) | 1 (1)
oozing around PICC line-blood (Vascular disorders) | 1 (1)
occasional cough and nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
ankle clonus (Nervous system disorders) | 2 (2)
increased patellar reflexes (Nervous system disorders) | 2 (2)
elevated alkaline phosphatase (Hepatobiliary disorders) | 1 (1)
bilirubin +1 in urine (Renal and urinary disorders) | 1 (1)
intermittent stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
decreased muscle tone in extremities (Nervous system disorders) | 1 (1)
diastasis recti (Musculoskeletal and connective tissue disorders) | 1 (1)
head lag (Nervous system disorders) | 1 (1)
Horner Syndrome (Nervous system disorders) | 1 (1)
increased hepatomegaly (Hepatobiliary disorders) | 1 (1)
increased splenomegaly (Hepatobiliary disorders) | 1 (1)
dacryostenosis, left eye (Eye disorders) | 1 (1)
increased GGT (Hepatobiliary disorders) | 1 (2)
Sandifer syndrome (Gastrointestinal disorders) | 1 (1)
increased AST (Hepatobiliary disorders) | 1 (1)
increased ALT (Hepatobiliary disorders) | 1 (1)
fever (Infections and infestations) | 1 (1)
viral exthanthem (Infections and infestations) | 1 (1)
hypernatremia (Metabolism and nutrition disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
increased BUN (Renal and urinary disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1)
platelet count decreased (Blood and lymphatic system disorders) | 1 (1)
hematuria (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT03471143/Prot_SAP_001.pdf